CLINICAL TRIAL: NCT03208231
Title: Phase I/II Multisite, Randomized, Controlled Study of Monoclonal Antibody VRC01 With Combination Antiretroviral Therapy to Promote Clearance of HIV-1-Infected Cells in Infants
Brief Title: Evaluating the Safety and Antiviral Activity of Monoclonal Antibody VRC01 in Infants With HIV Receiving Combination Antiretroviral Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2008; 20735 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VRC01 (Arm 1) (Experimental): Infants received VRC01 subcutaneous injections (40 mg/kg) at Weeks 0, 2, 6, and 10.
  Interventions: Biological: VRC01; Drug: Combination Antiretroviral Therapy (cART)
- No-VRC01 (Arm 2) (Active Comparator): Infants did not receive VRC01.
  Interventions: Drug: Combination Antiretroviral Therapy (cART)

INTERVENTIONS:
Biological: VRC01 — 40 mg/kg of VRC01 administered by subcutaneous injection.
  Other Names: VRC-HIVMAB060-00-AB
  Arms: VRC01 (Arm 1)
Drug: Combination Antiretroviral Therapy (cART) — All infants received non-study provided cART selected by their primary care provider and supplied through non-study sources (i.e., cART not provided through the study).

SUMMARY:
The purpose of this study was to evaluate the safety and antiviral activity to promote clearance of HIV-1 infected cells of VRC01 in infants with HIV beginning combination antiretroviral therapy (cART).

DETAILED DESCRIPTION:
VRC01 is an experimental human immunoglobulin G1 (IgG1) monoclonal antibody. The purpose of this study was to evaluate the safety and antiviral activity to promote clearance of HIV-1 infected cells of VRC01 received within 12 weeks of birth in infants with HIV initiating cART.

All infants were required to have initiated cART within 14 days before or at study entry. Infants were randomly assigned to either receive VRC01 (VRC01, Arm 1) or not receive VRC01 (No-VRC01, Arm 2). Randomization was stratified by whether the initial cART regimen included an integrase inhibitor.

Infants in the VRC01 arm received VRC01 injections at study entry (Week 0) and Weeks 2, 6, and 10. Infants in the No-VRC01 arm received no study product.

Infants attended study visits at Weeks 1, 2, 3, 6, 7, 10, 11, 14, 16, 20, 24, 36, and 48. Visits included physical examinations, blood and urine collection.

Infants' mothers could optionally be enrolled in the study for one-time specimen collection for exploratory evaluations. Maternal study participation was not required for infant study participation.

The study was closed to enrollment prematurely on March 19, 2020 due to the outbreak of coronavirus disease 2019 (COVID-19) and after enrolling 61 of the targeted 68 infants.

ELIGIBILITY:
Infant Inclusion Criteria:

* Weigh at least 2500 grams
* Confirmed HIV-1 infection
* The following laboratory values at screening:

  * Cluster of differentiation 4 (CD4) lymphocyte percentage greater than 15
  * Severity grade 1 or lower hemoglobin, platelet count, and absolute neutrophil count
  * Severity grade 1 or lower alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase
* First dose of initial combination antiretroviral therapy (cART) regimen taken on the day of randomization or within 14 days prior to the day of randomization
* Expected to be available for 48 weeks of follow-up at study entry
* Parent or legal guardian willing and able to provide written informed consent for infant participation in the study
* Parent or legal guardian willing and able to complete reactogenicity memory aids for study purposes, based on parent/guardian report.

Infant Exclusion Criteria:

* Infant or infant's mother received exclusionary active or passive HIV-specific immunotherapy
* Initiated a combination of three or more antiretrovirals, all at or above recommended treatment doses, within 48 hours of birth
* Received within 30 days prior to study entry, or was identified as requiring, any of the following:

  * Chronic (more than 14 days) systemic steroid treatment
  * Immunoglobulin treatment
  * Immunomodulators (interleukins, interferons, cyclosporin)
  * Cytotoxic chemotherapy
  * Treatment for active tuberculosis (TB) disease
  * Any investigational agent
  * Note: Treatment for latent TB infection was permitted
* Any documented or suspected clinically significant medical illness, clinically significant congenital anomaly, or immediately life-threatening condition that, in the opinion of the site investigator or designee, would interfere with the infant's ability to comply with study requirements
* Any other condition that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Maternal Inclusion Criteria (maternal study participation was not required for infant study participation):

The mothers of enrolled infants were asked to consent to blood collection and storage for this study. The following criteria must have been met in order for mothers to undergo blood collection for this purpose:

* Mother was willing and able to provide independent written informed consent for blood collection and storage for virology and immunology investigations
* Mother had no documented or suspected condition that, in the opinion of the site investigator or designee, would make blood collection unsafe

Ages: 0 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth (Betsy) McFarland, MD, Study Chair — University of Colorado School of Medicine; Alka Khaitan, MD, Study Chair — Indiana University School of Medicine
Locations (7):
- Botswana (2):
  - Molepolole CRS, Molepolole, Kweneng District
  - Gaborone CRS, Gaborone, South-East District
- Brazil (2):
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
- Malawi (2):
  - Malawi CRS, Lilongwe, Central Region
  - Blantyre CRS, Blantyre
- Harare Family Care CRS, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data."
URL: https://www.impaactnetwork.org/

REFERENCES:
- [Background] Khaitan A, Lindsey J, Capparelli E, Tierney C, Coletti A, Perlowski C, Cotton MF, Yin DE, Majji S, Moye J, Spiegel H, Harding P, Costello D, Krotje C, Gama L, Persaud D, McFarland EJ, on behalf of the IMPAACT 2008 Protocol Team. Phase I/II Study of monoclonal antibody VRC01 with early antiretroviral therapy to promote clearance of HIV-1 infected cells in infants (IMPAACT 2008). Oral presentation at 24th International AIDS Conference, July 2022.
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (AE) Grading Table, Corrected Version 2.1, dated July 2017. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events (EAE) to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 infants were enrolled at 7 sites in 4 countries (Botswana, Malawi, Zimbabwe and Brazil) between August 6, 2018 and March 11, 2020.
Pre-assignment Details: Infants were randomized equally to the two study arms. Randomization was stratified by whether their initial combination antiretroviral (cART) regimen included an integrase inhibitor.
Groups:
- VRC01 (Arm 1): Infants received VRC01 subcutaneous injections (40 mg/kg) at Weeks 0, 2, 6, and 10.
  All infants on cART.
- No-VRC01 (Arm 2): Infants did not receive VRC01.
  All infants on cART.
Period: Overall Study
Arm/Group | VRC01 (Arm 1) | No-VRC01 (Arm 2)
Started | 30 | 31
Evaluable (One infant in No-VRC01 arm did not return to the clinic after Week 0. This infant was not included in analyses of outcome measures.) | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 3
Not completed — Death | 1 | 2
Not completed — Moved and unable to get to clinic | 1 | 0
Not completed — Unwilling to adhere to study requirements | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRC01 (Arm 1) | No-VRC01 (Arm 2) | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: Days] | 72 [56 to 82] | 73 [65 to 82] | 73 [64 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 16 | 10 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Black Non-Hispanic | 25 | 26 | 51
  Race/ethnicity: Hispanic (Regardless of Race) | 5 | 5 | 10
Region of enrollment [Count of Participants; unit: Participants]
  Botswana | 0 | 7 | 7
  Brazil | 3 | 3 | 6
  Malawi | 25 | 17 | 42
  Zimbabwe | 2 | 4 | 6
Days on antiretrovirals prior to study entry [Median (Full Range); unit: Days] | 8 [0 to 14] | 6 [0 to 13] | 7 [0 to 14]
Days on antiretrovirals prior to study entry [Count of Participants; unit: Participants]
  0 | 1 | 5 | 6
  1-7 | 11 | 15 | 26
  >7 | 18 | 11 | 29
HIV-1 RNA (copies/ml) [Count of Participants; unit: Participants]
  <1000 copies/ml | 2 | 3 | 5
  1000 - < 10,000 copies/ml | 10 | 8 | 18
  10,000 - < 100,000 copies/ml | 11 | 10 | 21
  >= 100,000 copies/ml | 7 | 10 | 17
HIV-1 RNA (copies/ml) [Median (Inter-Quartile Range); unit: copies/ml] | 12,552 [5,050 to 95,395] | 22,625 [3,360 to 523,120] | 16,566 [4,290 to 117,165]
HIV-1 DNA (log10 copies/million PBMCs) [Median (Inter-Quartile Range); unit: log10 copies/million PBMCs] — Population: One infant in No-VRC01 arm did not return to the clinic after entry and their entry HIV-1 DNA was not included.
  log10 copies/million PBMCs
    number analyzed (Participants) | 30 | 30 | 60
    (all) | 3.12 [2.75 to 3.32] | 3.16 [2.75 to 3.46] | 3.15 [2.75 to 3.35]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants Experiencing at Least One Grade 3 or Higher Adverse Event (AE)
Description: Includes reactogenicity outcomes, abnormal laboratory test results, signs, symptoms, and diagnoses. Adverse event severity grading was based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Two-sided exact 95% Clopper-Pearson confidence intervals were calculated.
Time Frame: From Week 0 to Week 14
Population: One infant in the No-VRC01 arm did not return to clinic after Week 0 and is not included in the analysis population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VRC01 (Arm 1) | No-VRC01 (Arm 2)
Number analyzed (Participants) | 30 | 30
Percentage of participants | 40.0 [22.7 to 59.4] | 46.7 [28.3 to 65.7]
Statistical Analysis 1: Comparison: VRC01 (Arm 1) vs No-VRC01 (Arm 2); Test type: Superiority; p = 0.79, Fisher Exact

2. Primary Outcome: Change in HIV-1 DNA Concentration in Peripheral Blood Mononuclear Cells (PBMCs) From Week 0 to Week 14
Description: Mean changes (Week 14 - Week 0) were calculated on log10-transformed HIV-1 DNA concentration. Values below the assay detection limit were set to half the lower assay limit of 4.09 copies/million PBMCs. Values above the detection limit were set to the upper limit of 10,000 copies/million PBMCs.
Time Frame: Week 0 and Week 14
Population: One infant in No-VRC01 arm did not return to clinic after week 0 and is not included in analysis population
Measure: Median (Inter-Quartile Range); unit: log10 copies/million PBMCs
Arm/Group | VRC01 (Arm 1) | No-VRC01 (Arm 2)
Number analyzed (Participants) | 30 | 30
log10 copies/million PBMCs | -0.41 [-0.56 to -0.30] | -0.53 [-0.70 to -0.33]
Statistical Analysis 1: Comparison: VRC01 (Arm 1) vs No-VRC01 (Arm 2); Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Median Pre-dose VRC01 Concentrations in the Plasma (VRC01 Arm Only)
Description: Median (mcg/ml) pre-dose VRC01 concentrations in the plasma (VRC01 Arm only)
Time Frame: Weeks 2, 6, 10, 14, and 16
Population: One infant had no PK measurements run as sample sent to incorrect location for testing.
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | VRC01 (Arm 1)
Number analyzed (Participants) | 29
mcg/ml
  Week 2 | 109.4 [91.3 to 132.1]
  Week 6 | 79.5 [52.9 to 114.5]
  Week 10 | 96.5 [38.5 to 113.3]
  Week 14 | 82.3 [27.0 to 105.9]
  Week 16 | 53.2 [15.5 to 78.6]

4. Secondary Outcome: Geometric Mean of Pre-dose VRC01 Concentrations in the Plasma (VRC01 Arm Only)
Description: Geometric mean (mcg/ml) of pre-dose VRC01 concentrations with 90% confidence intervals
Time Frame: Weeks 2, 6, 10, 14, and 16
Population: One infant had no PK measurements run as sample sent to incorrect location for testing.
Measure: Geometric Mean (90% Confidence Interval); unit: mcg/ml
Arm/Group | VRC01 (Arm 1)
Number analyzed (Participants) | 29
mcg/ml
  Week 2: number analyzed (Participants) | 28
  Week 2 | 104.2 [90.1 to 120.4]
  Week 6: number analyzed (Participants) | 28
  Week 6 | 64.7 [45.8 to 91.4]
  Week 10: number analyzed (Participants) | 28
  Week 10 | 57.5 [35.7 to 92.5]
  Week 14 | 47.6 [29.0 to 78.1]
  Week 16: number analyzed (Participants) | 28
  Week 16 | 26.7 [14.8 to 48.4]

5. Secondary Outcome: Percentage of Infants With Pre-dose VRC01 Concentrations >= 20 mcg/ml in the Plasma (VRC01 Arm Only)
Description: Percentage of infants with pre-dose VRC01 concentrations >= 20 mcg/ml in the plasma (VRC01 Arm only)
Time Frame: Weeks 2, 6, 10, 14, 16
Population: One infant had no PK measurements run as sample sent to incorrect location for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 (Arm 1)
Number analyzed (Participants) | 29
Participants
  Week 2: number analyzed (Participants) | 28
  Week 2 | 28
  Week 6: number analyzed (Participants) | 28
  Week 6 | 25
  Week 10: number analyzed (Participants) | 28
  Week 10 | 25
  Week 14 | 24
  Week 16: number analyzed (Participants) | 28
  Week 16 | 18

6. Secondary Outcome: Percentage of Infants With Pre-dose VRC01 Concentrations >= 50 mcg/ml in the Plasma (VRC01 Arm Only)
Description: Percentage of infants with pre-dose VRC01 concentrations >= 50 mcg/ml in the plasma (VRC01 Arm only)
Time Frame: Weeks 2, 6, 10, 14, 16
Population: One infant had no PK measurements run as sample sent to incorrect location for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 (Arm 1)
Number analyzed (Participants) | 29
Participants
  Week 2: number analyzed (Participants) | 28
  Week 2 | 27
  Week 6: number analyzed (Participants) | 28
  Week 6 | 21
  Week 10: number analyzed (Participants) | 28
  Week 10 | 20
  Week 14 | 18
  Week 16: number analyzed (Participants) | 28
  Week 16 | 15

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Week 48 or premature study discontinuation.
Description: Complete blood count and selected chemistries assessed at screening, Weeks 1, 3, 7, 11, 14, 20, and 24. Signs, symptoms and diagnoses were recorded up to Week 16 if >= Grade 1 and after Week 16 if >= Grade 2. AE severity was graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 except for axillary measured fever and injection site pain/tenderness, which were graded according to study-specific criteria in Section 7.3.3 of the Protocol.
Groups:
- VRC01: Infants received VRC01 subcutaneous injections (40 mg/kg) at Weeks 0, 2, 6, and 10.
  All infants on cART.
- No-VRC01: Infants did not receive VRC01.
  All infants on cART.
Arm/Group | VRC01 | No-VRC01
All-Cause Mortality (participants affected / at risk) | 1/30 | 2/30
Serious Adverse Events (participants affected / at risk) | 7/30 | 11/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VRC01 (N=30) | No-VRC01 (N=30)
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Otitis media (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Infantile vomiting (Gastrointestinal disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Plasmodium falciparum infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VRC01 (N=30) | No-VRC01 (N=30)
Anaemia (Blood and lymphatic system disorders) | 15 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 1
Otorrhoea (Ear and labyrinth disorders) | 2 | 1
Eye discharge (Eye disorders) | 0 | 2
Lid sulcus deepened (Eye disorders) | 1 | 2
Ocular hyperaemia (Eye disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 10
Infantile vomiting (Gastrointestinal disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 6 | 1
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 10 | 9
Vaccination site induration (General disorders) | 2 | 0
Acarodermatitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 4 | 3
Folliculitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 6 | 7
Oral candidiasis (Infections and infestations) | 4 | 4
Otitis media acute (Infections and infestations) | 5 | 4
Pharyngitis (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pyuria (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 5
Urinary tract infection (Infections and infestations) | 4 | 3
Alanine aminotransferase increased (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 9
Blood creatinine increased (Investigations) | 0 | 2
Blood potassium increased (Investigations) | 2 | 0
Breath sounds abnormal (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 27 | 28
Neutrophil count decreased (Investigations) | 21 | 15
Platelet count decreased (Investigations) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Poor feeding infant (Metabolism and nutrition disorders) | 2 | 1
Underweight (Metabolism and nutrition disorders) | 2 | 1
Infant irritability (Nervous system disorders) | 3 | 0
Irritability (Psychiatric disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 2
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 2
Papule (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Accrual into the study was terminated early due to the outbreak of coronavirus disease 2019 (COVID-19), with 60 evaluable infants out of the targeted 68.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (7):
  • Study Protocol: Protocol Version 2.0 (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/Prot_001.pdf
  • Study Protocol: Letter of Amendment 1.0 (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/Prot_002.pdf
  • Study Protocol: Letter of Amendment 2.0 (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/Prot_003.pdf
  • Study Protocol: Protocol Clarification Memo 1.0 (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/Prot_004.pdf
  • Study Protocol: Protocol Clarification Memo 2.0 (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/Prot_005.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/SAP_006.pdf
  • Informed Consent Form (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03208231/ICF_000.pdf